CLINICAL TRIAL: NCT04423562
Title: Investigation of the Prognostic Value of pVO2 in Recipients of Left Ventricular Assist Devices
Brief Title: PROgnostic Value of Exercise Capacity Measured as Peak Oxygen Uptake (pVO2) in Recipients of Left Ventricular Assist Devices
Acronym: PRO-VAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Finn Gustafsson, Professor, Rigshospitalet, Denmark
Other Study IDs: 330131365/2
Record Dates: First submitted 2020-05-03; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Left Ventricular Assist Device; Prognosis; Advanced Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Durable LVAD recipient with post implant VO2
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Pooling of earlier VO2-studies conducted at the dept. of cardiology, Rigshospitalet, Denmark, and all LVAD centres of the World that wish to participate.

The purpose is to investigate the prognostic value of VO2 in recipients of durable LVADs using data from studies already conducted.

DETAILED DESCRIPTION:
Background and purpose:

Peak oxygen uptake (pVO2) is used extensively in HF to predict prognosis and time for heart transplantation. Many centers are increasingly measuring pVO2 in LVAD supported HF patients, though this has mostly been for research or rehabilitation purposes. It is unknown if pVO2 predicts outcome in LVAD treated HF patients.

The investigators will pool data from all willing centers of the World to investigate the prognostic value of pVO2 (e.g. outcome in LVAD supported patients) and, secondly the investigators will investigate wether the predictive power of pVO2 in LVAD recipients depends on the treatment indication (BTT and DT).

Methods:

Data is collected in anonymized form from all centers willing to contribute data.

Hypothesis:

The hypothesis is that lower pVO2 is associated with higher rates of death or urgent transplantation (primary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Durable LVAD implantation
* VO2 in stable post implant phase

Exclusion Criteria:

* No VO2 data available
* Concomittant RVAD (temp/durable device)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients implanted with a durable LVAD (post-2006) and available post implant VO2 (stable phase) can be included in this study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Outcome after implantation | Stable-phase post implant VO2 (e.g. >3months and up to 13 year post implant)
  Survival/ongiong on device/explant/htx after LVAD implantation

CONTACTS AND LOCATIONS:
Overall Officials: Finn Gustafsson, MD,PhD,DMSci, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, DK, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mirza KK, Szymanski MK, Schmidt T, de Jonge N, Brahmbhatt DH, Billia F, Hsu S, MacGowan GA, Jakovljevic DG, Agostoni P, Trombara F, Jorde U, Rochlani Y, Vandersmissen K, Reiss N, Russell SD, Meyns B, Gustafsson F; PRO-VAD Investigators. Prognostic Value of Peak Oxygen Uptake in Patients Supported With Left Ventricular Assist Devices (PRO-VAD). JACC Heart Fail. 2021 Oct;9(10):758-767. doi: 10.1016/j.jchf.2021.05.021. Epub 2021 Aug 11. PMID 34391745